CLINICAL TRIAL: NCT05379569
Title: Shanghai General Hospital, Shanghai, Jiao Tong University School of Medicine
Brief Title: Comparative Study of BFC and BuCy Conditioning Regimen for Allo-PBSCT in Acute B-cell ALL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Department of Hematology，Director, Head of Otolaryngology, Principal Investigator,, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-B-ALL
Record Dates: First submitted 2022-05-03; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Acute B Lymphoblastic Leukemia; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conditioning regimen with Malilane,cyclophosphamide and fludarabine (Experimental): Malilane 3.2mg/kg/d *4d (-5,-4,-3,-2day) cyclophosphamide 25mg/kg/d*4d (-9-8,-7,-6 day) fludarabine 30mg/m2/d*4d (-9-8,-7,-6 day) Donor stem cells will be transfused at 0 days.
  Interventions: Drug: Fludarabine
- conditioning regimen with Malilane and cyclophosphamide (Active Comparator): malilane 3.2mg/kg *4d (-5,-4,-3,-2day) cyclophosphamide 50mg/kg/d*2d (-2,-1day) Donor stem cells will be transfused at 0 days.
  Interventions: Drug: Fludarabine

INTERVENTIONS:
Drug: Fludarabine — The combination of fludarabine and cyclophosphamide has synergistic effect, which can better kill B lymphocyte, and can enhance the killing effect of pretreatment regimen on B lymphocyte tumor.
  Other Names: Malilane and cyclophosphamide

SUMMARY:
Comparing the efficacy and safety of fludarabine-containing BFC conditioning regimen with traditional BuCy conditioning regimen in Acute B-cell lymphoblastic leukemia patients who treated with allogeneic hematopoietic stem cell transplantation, to establish a conditioning regimen for improving the survival rate of patients with B-cell ALL after transplantation.

Acute B-cell lymphoblastic leukemia (B-ALL) is a hematologic malignancy . The incidence of B-All is higher in children than in adults, but more than 80% of children patients can be cured by chemotherapy, while the survival rate of adult patients is less than 40%. Recurrence or progression of the disease is the main reason affecting the survival of patients.

Although CD19-targeted CAR T cell therapy is an effective salvage treatment for relapsed and refractory B-ALL, bridging allogeneic hematopoietic stem cell transplantation is required after remission. 1-year LFS and 1-year OS were 11.6% and 32% in patients without bridging grafts after CAR T.

Allogeneic hematopoietic stem cell transplantation is an effective treatment for ALL. Before the transplant, patients receive high doses of chemotherapy plus or total body irradiation（TBI） to 'creation of space' ，immunosuppression and disease eradication. This is called conditioning regimen. Conditioning regimen plays a key role in reducing tumor load and diseaseconditioning regimen recurrence.

Conditioning regimen for different diseases are different. Conditioning regimen are based on TBI and chemotherapy BuCy, with low TBI recurrence rate but high treatment-related mortality (TRM). BuCY chemotherapy had low TRM but high recurrence rate, so there was no difference in total OS. Therefore, it is of great clinical value to explore a conditioning regimenprogram. How to optimize the preconditioning program before transplantation, so as to reduce the recurrence rate and prolong the survival period of adult B-cell ALL patients after transplantation has become a issue that needs to be solved urgently in clinical practice.

BFC (Malilane + fludarabine + cyclophosphamide) is the addition of fludarabine to BuCy (malilane + cyclophosphamide). The combination of fludarabine and cyclophosphamide has synergistic effect, which can better kill B lymphocyte, and can enhance the killing effect of pretreatment regimen on B lymphocyte tumor.

DETAILED DESCRIPTION:
This study was a prospective, randomized, controlled, single-center clinical study. A total of 142 patients eligible for the inclusion of acute B lymphoblastic leukemia were randomly divided into two groups: the experimental group (n = 71) and the control group (n = 71). The treatment group was given BFC conditioning regimen (fludalabine, marylan, cyclophosphamide), and the control group was given BuCY conditioning regimen (marylan, cyclophosphamide), and the patients were followed up to 1 year after transplantation. The 1-year disease-free survival rate of patients in the two groups was compared to evaluate whether increasing fludarabine could reduce the recurrence rate of patients after transplantation and thus improve the overall survival rate.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-55.
2. The patient was diagnosed as acute B-lymphoblastic leukemia, which was confirmed by bone marrow cell morphology, cytochemistry, immunotyping and chromosome examination, including acute chronic myelocytic leukemia, Ph-acute B-lymphoblastic leukemia, and acute B-lymphoblastic leukemia after CART treatment.
3. The diagnostic criteria for b-blastic leukemia in remission were: complete hematologic response (CR) with negative minimal residual lesions (MRD) after regular induction of remission chemotherapy, or complete hematologic response with negative MRD after CART treatment.
4. ECOG physical fitness status score ≤2.
5. All organs function normally and meet the following inspection standards:

   A) Liver function ALT, AST and TBIL≤2 times the upper limit of normal value B) BUN and Cr of renal function ≤1.25 times the upper limit of normal value.
6. Have the following cardiac function conditions: ecg examination did not indicate any acute myocardial infarction, arrhythmia or atrioventricular block of degree I or above; Centerless incomplete function; No active rheumatic heart disease; There was no indication of cardiac enlargement on chest radiograph or physical examination.

(7) The patient had a qualified allogeneic hematopoietic stem cell transplantation donor, including haploid, myeloma and sibling.

8) The patient and its legal client have the desire and requirement for hematopoietic stem cell transplantation, and sign the informed consent, and are willing to and abide by the treatment plan, follow-up plan, laboratory examination, etc.

9) The donor meets the donation requirements-

Exclusion Criteria:

1. There are any contraindications for allogeneic hematopoietic stem cell transplantation.
2. Ph+ acute lymphoblastic leukemia
3. Serious damage of important organ functions, such as respiratory failure, heart failure, decompensated liver insufficiency, renal insufficiency, etc.
4. Pregnant or lactating women.
5. Those who are undergoing clinical trials of other drugs.
6. Patients suffering from other serious acute or chronic physical or mental diseases, or abnormal laboratory examination, which may affect the administration of study drugs and the researchers' judgment of the condition and interpretation of the test results, are not suitable to participate in the clinical trial.
7. The donor does not fit the conditions of the donor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
RFS | one year
  Relapse-free survival

SECONDARY OUTCOMES:
OS (OS). | one year
  overall survival
RR | one year
  relapse rate
AE | one year
  adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No